CLINICAL TRIAL: NCT00001083
Title: A Phase II Rolling Arm Master Protocol (PRAM) of Novel Antiretroviral Therapy in Stable Experienced HIV- Infected Children; PRAM-1: ZDV+3TC vs. d4T+Ritonavir vs. ZDV+3TC+Ritonavir; PRAM-1, Step 2: d4T+Nevirapine+Ritonavir; PRAM-1, Step 3: d4T+Indinavir vs. ZDV+3TC+Indinavir
Brief Title: Comparison of New Anti-HIV Drug Combinations in HIV-Infected Children Who Have Taken Anti-HIV Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 338; 11309 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Zidovudine; Nevirapine; Stavudine; HIV Protease Inhibitors; Ritonavir; Lamivudine; Indinavir; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir; Nevirapine; Lamivudine; Stavudine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir
Drug: Nevirapine
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
For PRAM-1: To evaluate zidovudine (ZDV) + lamivudine (3TC) vs. stavudine (d4T) + ritonavir vs. ZDV + 3TC + ritonavir with respect to the change in plasma HIV-1 RNA copy number from baseline to 48 weeks [AS PER AMENDMENT 1/5/98: 72 weeks; AS PER AMENDMENT 7/17/98: 48 weeks] in stable HIV-infected children with >= 16 weeks of prior continuous antiretroviral therapy. To evaluate the safety and tolerance of ZDV + 3TC vs. d4T + ritonavir vs. ZDV + 3TC + ritonavir based upon laboratory and clinical toxicities.

AS PER AMENDMENT 10/20/97: For PRAM-1, Step 2: To evaluate d4T + nevirapine + ritonavir with respect to change in plasma HIV-1 RNA copy number from baseline to 48 weeks in children who have received at least 12 weeks of therapy on the PRAM-1 ZDV/3TC arm and have over 10,000 viral copies at weeks 12, 24, or 36. To evaluate the safety and tolerance of d4T + nevirapine + ritonavir based upon laboratory and clinical toxicities. [AS PER AMENDMENT 10/23/98: To evaluate safety and tolerance of a switch from d4T + ritonavir vs. ZDV + 3TC + ritonavir to d4T + indinavir vs. ZDV + 3TC + indinavir in stable, HIV-infected children with RNA values <= 10,000 copies/ml.] For PRAM-1: Evidence supports combination therapy with 2 or more antiviral agents as beneficial in the long-term management of HIV. The possibility exists that combination therapy may result in a synergistic or additive activity over a prolonged period of time. Also hypothesized is that the development of resistance to individual agents will be developed if viral replication is significantly decreased.

AS PER AMENDMENT 10/20/97: For PRAM-1, Step 2: Interim analysis at 12 weeks on PRAM-1 indicates that the proportion of children reaching undetectable RNA levels on the ZDV + 3TC arm is significantly less than the other two arms. The protocol, therefore, has been modified (Step 2) to permit children in the ZDV + 3TC arm with RNA copy number >= 10,000 the opportunity to change to a novel therapeutic regimen (d4T + nevirapine + ritonavir).

DETAILED DESCRIPTION:
For PRAM-1: Evidence supports combination therapy with 2 or more antiviral agents as beneficial in the long-term management of HIV. The possibility exists that combination therapy may result in a synergistic or additive activity over a prolonged period of time. Also hypothesized is that the development of resistance to individual agents will be developed if viral replication is significantly decreased.

AS PER AMENDMENT 10/20/97: For PRAM-1, Step 2: Interim analysis at 12 weeks on PRAM-1 indicates that the proportion of children reaching undetectable RNA levels on the ZDV + 3TC arm is significantly less than the other two arms. The protocol, therefore, has been modified (Step 2) to permit children in the ZDV + 3TC arm with RNA copy number >= 10,000 the opportunity to change to a novel therapeutic regimen (d4T + nevirapine + ritonavir).

The Master PRAM is a Phase II, multicenter, randomized, open-label trial of a standard therapeutic regimen in current use versus experimental therapies administered over 48 weeks. It is designed to allow new therapeutic arms to be studied as "rolling screens" through multiple generations of PRAM. Each PRAM generation compares 2 novel therapeutic arms with a linking arm that allows for an indirect comparison of included therapies. Once accrual to PRAM-1 is complete a new treatment comparison opens for accrual (PRAM-2). The linking arm to be used in PRAM-2 is decided by the Pediatric Primary Scientific Committee. PRAM-2 will continue to accrue patients while PRAM-1 patients continue therapy.

For PRAM-1: This study compares the following three treatment arms:

Arm I: ZDV plus 3TC Arm II: d4T plus ritonavir Arm III: ZDV plus 3TC plus ritonavir. Prior to randomization to one of the three arms, patients are stratified based on CD4 percents: either less than 15% or greater than or equal to 15%. The first 8 patients randomized to Arms II and III participate in a real-time Phase I pharmacokinetic study (16 patients total). After the first 45 (15 per arm) patients entered are followed for 24 weeks, an interim analysis is done. Patients are treated for 48 weeks [AS PER AMENDMENT 1/5/98: 72 weeks].

AS PER AMENDMENT 10/20/97:

PRAM-1, Step 2:

Patients initially assigned to Arm I (ZDV plus 3TC) who have RNA values greater than 10,000 copies at week 12, 24, or 36 are assigned to switch protocol treatment to d4T + ritonavir + nevirapine. Patients may enroll in Step 2 no later than week 38 of PRAM-1. [AS PER AMENDMENT 1/5/98: Patients initially assigned to Arm 1 with viral load greater than 100,000 copies may also switch to Step 2 or discontinue therapy. Patients originally assigned to Arms I or II with viral load greater than 10,000 may continue their current drugs or discontinue study therapy; those with viral load greater than 100,000 should discontinue study drugs.] [AS PER AMENDMENT 7/17/98: PRAM-1 has been extended to permit long-term follow-up of clinically stable, HIV-infected children for a total of 120 weeks. Patients still on initial treatment assignment for all three treatment arms are eligible for this extension, as are children from PRAM-1, Step 2. Step 2 is now closed to enrollment. Patients on 3TC/ZDV who reach virologic failure must discontinue study therapy].

[AS PER AMENDMENT 10/23/98: PRAM-1, Step 3: This amendment substitutes indinavir (IDV) capsules for ritonavir capsules in PRAM-1. The regimens will switch from d4T plus ritonavir versus ZDV plus 3TC plus ritonavir to d4T plus IDV versus ZDV plus 3TC plus IDV. All patients will be followed for 48 weeks. Patients eligible for this change in regimens are those taking ritonavir capsules who have RNA values less than or equal to 10,000 copies/ml (as demonstrated by the most recent viral load test) after at least 72 weeks on PRAM-1, Step I. Twelve patients with RNA values less than or equal to 400 copies/ml will immediately join the study; 6 will receive d4T plus IDV and 6 will receive ZDV plus 3TC plus IDV. Additional patients may be added based on toxicity and viral load results. A total sample size of 53 evaluable patients (37 with RNA values less than or equal to 400 copies/ml and 16 with RNA values of greater than 400 to 10,000 copies/ml) is anticipated. PRAM-1 Step 2 patients are not eligible for Step 3. PRAM-1, Step 2 patients currently taking liquid ritonavir should continue their study drug; those taking ritonavir capsules will switch to liquid ritonavir or go off study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* IVIG and opportunistic infection prophylaxis will be allowed.
* Erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF) and granulocyte-macrophage colony- stimulating factor (GM-CSF) will be allowed for the management of hematologic toxicity.
* Treatment with trimethoprim is allowed at the discretion of the principal investigator.

Patients must have:

* Laboratory evidence (at least 2 viral tests) of HIV-1 infection.
* Clinical and immunological stability [maintained CDC category 1 or 2 immunologic status for past 4 months and no new CDC category (diagnosis within the past year)].
* Patients must have received continuous antiretroviral therapy for the past 16 weeks (missing no more than 6 weeks of therapy during the previous 16 weeks).

AS PER AMENDMENT 10/20/97: For PRAM-1, Step 2:

* Viral load >= 10,000 and < 100,000 copies/ml at week 12, 24, or 36 in children initially assigned to Arm I (ZDV + 3TC) of PRAM-1 and currently on study.

Prior Medication:

Required:

* Patients must have received continuous antiretroviral therapy for the past 16 weeks.

Allowed:

* Patients who have received immunomodulator therapy as part of perinatal clinical trials or in trials for HIV- exposed infants are eligible.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Current grade 3/4 clinical or laboratory toxicity and/or current grade 2 or higher amylase/lipase toxicity.
* Active opportunistic infection and/or serious bacterial infection.
* Current diagnosis of malignancy.

Concurrent Medication:

Excluded:

* Current antiretroviral therapy identical to any of the following regimens:
* ZDV + 3TC, d4T + ritonavir and ZDV + 3TC + ritonavir.
* Concurrent therapy with any other anti-HIV-1 therapy, biologic response modifiers (EPO, G-CSF and GM-CSF allowed), human growth hormone and megestrol acetate.
* Use of continuous systemic corticosteroids (>= 14 days duration) is not allowed.
* Medications that are incompatible with ritonavir.
* Probenecid and daily intravenous pentamidine.

[AS PER AMENDMENT 10/23/98: The following are excluded in patients receiving indinavir:

* terfenadine, astemizole, cisapride, rifampin, rifabutin, triazolam, ketoconazole, clarithromycin, carbamazepine, phenobarbital, phenytoin, calcium channel blockers, midazolam, and ergot derivatives.]

Patients with the following prior conditions and symptoms are excluded:

* Documented hypersensitivity to a therapy included in any of the treatment arms.

Prior Medication:

Excluded:

Investigational drug therapy within 2 weeks prior to randomization.

NOTE:

* Co-enrollment in ACTG 219, ACTG 220 and certain ACTG opportunistic infection protocols is allowed.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240
Dates: Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nachman S, Study Chair; Wiznia A, Study Chair
Locations (61):
- United States (58):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Univ of Connecticut / Farmington, Farmington, Connecticut
  - Yale Univ Med School, New Haven, Connecticut
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Florida Gainesville, Gainesville, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Palm Beach County Health Dept, Riviera Beach, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - UMDNJ - Robert Wood Johnson Med School / Pediatrics, New Brunswick, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - King's County Hosp Ctr / Pediatrics, Brooklyn, New York
  - SUNY - Brooklyn, Brooklyn, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Westchester Hosp, Valhalla, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Columbus Children's Hosp, Columbus, Ohio
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Med College of Virginia, Richmond, Virginia
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Result] Nachman S. Lack of improvement in growth in HIV-infected children on HAART 39th Intersci Conf Antimicrob Agents Chemother. 1999 Sept 26-29 (abstract no 120)
- [Result] Yogev R, Lee S, Wiznia A, Nachman S, Stanley K, Pelton S, Mofenson L, Fiscus S, Jimenez E, Rathore MH, Smith ME, Song LY, McIntosh K; Pediatrics AIDS Clinical Trials Group 338 Study Team. Stavudine, nevirapine and ritonavir in stable antiretroviral therapy-experienced children with human immunodeficiency virus infection. Pediatr Infect Dis J. 2002 Feb;21(2):119-25. doi: 10.1097/00006454-200202000-00007. PMID 11840078
- [Result] Nachman SA, Stanley K, Yogev R, Pelton S, Wiznia A, Lee S, Mofenson L, Fiscus S, Rathore M, Jimenez E, Borkowsky W, Pitt J, Smith ME, Wells B, McIntosh K. Nucleoside analogs plus ritonavir in stable antiretroviral therapy-experienced HIV-infected children: a randomized controlled trial. Pediatric AIDS Clinical Trials Group 338 Study Team. JAMA. 2000 Jan 26;283(4):492-8. doi: 10.1001/jama.283.4.492. PMID 10659875
- [Result] Nachman SA, Lindsey JC, Pelton S, Mofenson L, McIntosh K, Wiznia A, Stanley K, Yogev R. Growth in human immunodeficiency virus-infected children receiving ritonavir-containing antiretroviral therapy. Arch Pediatr Adolesc Med. 2002 May;156(5):497-503. doi: 10.1001/archpedi.156.5.497. PMID 11980557
- [Result] Jeremy RJ, Kim S, Nozyce M, Nachman S, McIntosh K, Pelton SI, Yogev R, Wiznia A, Johnson GM, Krogstad P, Stanley K; Pediatric AIDS Clinical Trials Group (PACTG) 338 & 377 Study Teams. Neuropsychological functioning and viral load in stable antiretroviral therapy-experienced HIV-infected children. Pediatrics. 2005 Feb;115(2):380-7. doi: 10.1542/peds.2004-1108. PMID 15687448
- [Result] Fiscus SA, Kovacs A, Petch LA, Hu C, Wiznia AA, Mofenson LM, Yogev R, McIntosh K, Pelton SI, Napravnik S, Stanley K, Nachman SA. Baseline resistance to nucleoside reverse transcriptase inhibitors fails to predict virologic response to combination therapy in children (PACTG 338). AIDS Res Ther. 2007 Feb 6;4:2. doi: 10.1186/1742-6405-4-2. PMID 17280617